CLINICAL TRIAL: NCT06754098
Title: An Off-Label Single Arm Clinical Study to Evaluate the Efficacy and Safety of Doxecitin and Doxribthymine in Adult Subjects With Thymidine Kinase 2 (TK2) Deficiency.
Brief Title: Doxecitin and Doxribthymine in Adult Subjects With Thymidine Kinase 2 (TK2) Deficiency
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cristina Domínguez González (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, Cristina Domínguez González, Doctor, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOTK2D; 2024-510763-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Thymidine Kinase 2 (TK2 ) Deficiency; Mitochondrial Myopathies
Keywords: TK2 deficiency; Primary Mitochondrial Myopathy; Deoxycytidine (dC); Deoxythymidine (dT); Mitochondrial DNA depletion and multiple deletions syndromes (MDDS)
MeSH Terms: conditions — Mitochondrial Myopathies

STUDY DESIGN:
Intervention Model Description: The study seeks to enroll 10 to 15 patients under follow-up in the Neuromuscular Unit of '12 de Octubre' Hospital. All subjects will be required to attend a screening visit at which their eligibility for the study will be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- doxecitin and doxribthymine (dT+dC) (Experimental): This is an open label study with all participants in a single arm. Study participants will take doxecitine and doxribtimine up to a maximum of 800 mg/kg/day (400 mg/kg/day doxecitine and 400 mg/kg/day doxiribtimine).
  Interventions: Drug: Doxecitine and Doxribtimine

INTERVENTIONS:
Drug: Doxecitine and Doxribtimine — A combination of doxecitine and doxribtimine is administered orally in 3 equal doses given approximately 6 to 8 hours apart .Dose will be increased if the tolerability profile is good.

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of Doxecitin and Doxribtimine (dC+dT) in adult participants with thymidine kinase 2 (TK2) deficiency attended in the Neuromuscular Unit of '12 de Octubre' Hospital.

The main questions it aims to answer are:

* Is dT+dC effective in the treatment of the adult participants with TK2 deficiency?
* Is dT+dC safe in the treatment of adult participants with TK2 deficiency?

Researchers will evaluate the effectiveness of the treatment doxecitin and doxribthymine in adult participants with TK2 deficiency. In addition, the mitochondrial DNA levels before and after treatment (extracted from the muscle and from uroepithelial cells) of these participants will be also studied.

DETAILED DESCRIPTION:
This is an Open Label, single-arm, single-center clinical study to evaluate the efficacy and safety of dT+dC in adults with TK2 deficiency (TK2d). TK2 deficiency is one of several mitochondrial autosomal recessive disorders that are collectively referred to as mitochondrial DNA depletion and multiple deletions syndromes (MDDS), in fact, TK2d is an ultra-rare disease, presenting as progressive proximal muscle weakness in all patients; however, clinical presentations are heterogeneous in nature and manifest with variable levels of severity and functional impairment across patients.

The study seeks to enroll patients under follow-up in the Neuromuscular Unit of '12 de Octubre' Hospital. All participants will be required to attend a screening visit at which their eligibility for the study will be determined. After signing the informed consent and verifying that they met all inclusion and exclusion criteria, participants will receive a daily dose of dT+dC in 3 equal divided doses administered orally at an approximate interval of 6 (±2) hours. dT+dC is to be initially dosed (commencing on Day 1) at 130 mg/kg/day of each nucleoside (130 mg/kg/day dC and 130 mg/kg/day dT), divided into 3 equal daily doses of approximately 43 mg/kg/dose. If the tolerability profile is acceptable after 2 weeks (approximately Day 15), the dose is to be increased to 260 mg/kg/day of each nucleoside (approximately 86 mg/kg/dose three-times daily, (TID). If the tolerability profile remains acceptable after an additional 2 weeks of dosing (approximately Day 29) the dose is to be further increased to 400 mg/kg/day (approximately 133 mg/kg/dose TID). The maximum dose is 400 mg/kg/day. The tolerability profile of the treatment will be evaluated based on whether the patient has diarrhea.

The total number of participants for the safety and efficacy analysis will be 10 to 15 participants with progressive myopathy with respiratory involvement.

The estimated duration of the study for individual participants will be 24 months. Although, based on previous experience in treating these patients, the investigators expect to see results within the first 6 to 12 months of treatment.

It is hypothesized that dT+dC oral administration is safe, well tolerated and clinically beneficial in adults with TK2 deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the subject.
2. Subject must be greater than 18 years of age at time of consent.
3. Genetic diagnosis of TK2 deficiency
4. Subject should have evidence of a moderate to severe disease, with motor and or respiratory involvement, shown by one of the following:

   1. North Star Ambulatory Assessment Scale (NSAA) less than 30
   2. 6-minute walking test less than 450 meters
   3. Force Vital Capacity in the sitting position less than 70 percent or a drop in the decubitus position greater than 10 percent or need for mechanical ventilation.
   4. Disabling symptoms and evidence of motor and/or respiratory function progressive decline.
5. Female subjects must have no intention to become pregnant during the study. Female subjects who are of childbearing potential (that is, following menarche until at least 1 year post-menopausal if not anatomically and physiologically incapable of becoming pregnant) must agree and commit to the use of highly effective methods of birth control for the duration of the study and for 30 days after the end of the study, and be willing to have additional pregnancy tests conducted during the study. Acceptable methods are defined as those that result, alone or in combination, in a low failure rate (that is, less than 1 percent per year) when used consistently and correctly, such as surgical sterilization, an intrauterine device, or hormonal contraception in combination with a barrier method.
6. Male subjects with partners of childbearing potential must agree to use effective contraception methods during the study and for at least 90 days after the last dose of the study medication. Acceptable methods include the use of condoms combined with spermicidal foam/gel/film/cream/suppository.
7. Willingness to comply with the study protocol, including but not limited to, all study procedures, study visits, and study drug compliance.

Exclusion Criteria:

1. History of liver disease, or liver function test results (alanine aminotransferase [ALT], aspartate transaminase [AST], or total bilirubin) greater than or equal2 times (2X) the upper limit of normal. Patients with transaminases greater than 2 times (2X) can participate with the approval and monitoring of a doctor specializing in liver toxicity.
2. Participation in a previous trial of any investigational agent for primary mitochondrial disease within 1 year prior to informed consent, or use of any other investigational therapy within 30 days (or 3 half-lives, whichever is longer) prior to informed consent, or participation in other clinical studies, within 30 days prior to informed consent, which in the opinion of the study Sponsor, may potentially confound results from this study.
3. Pregnant (females 10.0 years old or older will have a pregnancy test at screening), or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Motor Function Assessments: Neurological Exam using Medical Research Council (MRC Scale) Scale for Muscle Strength | Day 1, Months 1, 2, 3, 12, 15, 18, 21 and 24
  Motor Function will be measured using the MRC scale. The scale provides a measure of Muscle Strength across a range from 0 (No visible muscle contraction) to 5 (Full strength)
Efficacy - Motor Function Assessments: 6-minute walk test | Day 1, Months 1, 2, 3, 12, 15, 18, 21 and 24
  Motor Function will be measured using the 6-minute walk test (6MWT). Distance walked in meters over 6 minutes will be measured
Efficacy - Motor Function Assessments: North Star Ambulatory Assessment (NSAA) | Day 1, Months 1, 2, 3, 12, 15, 18, 21 and 24
  Motor function will be assessed using the NSAA scale. The NSAA is a 17-item scale that grades performance of various functional activities on a scale graded 0 (unable to complete the activity), 1 (completes the activity independently but with modifications), and 2 (completes the activity without modifications)
Efficacy - Motor Function Assessments: 100 meter-time velocity test | Day 1, Months 1, 2, 3, 12, 15, 18, 21 and 24
  Time to run 100 meters measured in seconds (sec)
Efficacy - Motor Function Assessments: Fatigue Scale test | Day 1, Months 1, 2, 3, 12, 15, 18, 21 and 24
  Motor function will be assessed Fatigue Scale test. The FACIT-Fatigue is a 13-item patient-reported outcome measure (range from 0 to 52: 0 = very much fatigued, 52 = not at all fatigued) assessing fatigue over the previous week
Efficacy - Respiratory Assessments measured by spirometry | Day 1, Months 1, 2, 3, 12, 15, 18, 21 and 24
  * Sitting Forced Vital Capacity (Sitting FVC) measure in percentage (%)
  * Drop in FVC lying down measured in percentage (%)
  * Maximal Inspiratory Pressure (MIP) measure in percentage: Evaluation of the strength of respiratory muscles is performed with measurements of MIP expressed in percentage (%)
  * Maximal Inspiratory Pressure (MEP) measure in percentage: Evaluation of the strength of respiratory muscles is performed with measurements of MEP expressed in percentage (%)
Efficacy - Respiratory Assessments: Use of ventilatory support (Use and Type ) | Day 1, Months 1, 2, 3, 12, 15, 18, 21 and 24
  Use and Type of mechanical ventilation (MV) [bilevel positive airway pressure (BiPAP) and/or continuous positive airway pressure (CPAP)] per subject will be assessed
Efficacy - Respiratory Assessments: Time of use of ventilatory support | Day 1, Months 1, 2, 3, 12, 15, 18, 21 and 24
  Total of hours of use of mechanical ventilation (MV) per subject will be assessed
Serum Biomarkers: lactate levels | Up to 24 months
  Number of participants with normal vs abnormal lactate levels measured in mmol/l
Serum Biomarkers: Growth/differentiation factor-15 (GDF15 ) | Up to 24 months
  Number of participants with normal vs abnormal Growth/differentiation factor-15 (GDF15) levels measured in mmol/l compared to normal ranges

SECONDARY OUTCOMES:
Safety as adverse events (AEs) | Up to 24 months
  Number of participants who experience adverse events (AEs)
Safety as serious adverse events (SAEs)adverse events | Up to 24 months
  Number of participants who experience serious adverse events (SAEs)

OTHER OUTCOMES:
Changes in the mtDNA levels before and after treatment | 6 month
  To assess change in mitochondrial DNA (mtDNA) levels, a muscle biopsy with a needle will be performed before entering the study and 6 months after the start of treatment
Changes in the peak oxygen consumption (VO2 max) test | 6 month
  A progressive exercise test will be undertaken at screening to assess peak oxygen consumption (VO2 max) using an electronically braked recumbent cycle ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina D Domínguez González, Dra., Principal Investigator — Hospital 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominguez-Gonzalez C, Badosa C, Madruga-Garrido M, Marti I, Paradas C, Ortez C, Diaz-Manera J, Berardo A, Alonso-Perez J, Trifunov S, Cuadras D, Kalko SG, Blazquez-Bermejo C, Camara Y, Marti R, Mavillard F, Martin MA, Montoya J, Ruiz-Pesini E, Villarroya J, Montero R, Villarroya F, Artuch R, Hirano M, Nascimento A, Jimenez-Mallebrera C. Growth Differentiation Factor 15 is a potential biomarker of therapeutic response for TK2 deficient myopathy. Sci Rep. 2020 Jun 22;10(1):10111. doi: 10.1038/s41598-020-66940-8. PMID 32572108
- [Background] Berardo A, Dominguez-Gonzalez C, Engelstad K, Hirano M. Advances in Thymidine Kinase 2 Deficiency: Clinical Aspects, Translational Progress, and Emerging Therapies. J Neuromuscul Dis. 2022;9(2):225-235. doi: 10.3233/JND-210786. PMID 35094997
- [Background] Bermejo-Guerrero L, Hernandez-Voth A, Serrano-Lorenzo P, Blazquez A, Martin-Jimenez P, Martin MA, Dominguez-Gonzalez C. Remarkable clinical improvement with oral nucleoside treatment in a patient with adult-onset TK2 deficiency: A case report. Mitochondrion. 2024 May;76:101879. doi: 10.1016/j.mito.2024.101879. Epub 2024 Apr 9. PMID 38599303
- [Background] Dominguez-Gonzalez C, Madruga-Garrido M, Mavillard F, Garone C, Aguirre-Rodriguez FJ, Donati MA, Kleinsteuber K, Marti I, Martin-Hernandez E, Morealejo-Aycinena JP, Munell F, Nascimento A, Kalko SG, Sardina MD, Alvarez Del Vayo C, Serrano O, Long Y, Tu Y, Levin B, Thompson JLP, Engelstad K, Uddin J, Torres-Torronteras J, Jimenez-Mallebrera C, Marti R, Paradas C, Hirano M. Deoxynucleoside Therapy for Thymidine Kinase 2-Deficient Myopathy. Ann Neurol. 2019 Aug;86(2):293-303. doi: 10.1002/ana.25506. Epub 2019 Jun 17. PMID 31125140